CLINICAL TRIAL: NCT02661217
Title: A Multicenter, Randomized, Open Label, Parallel Group Study Comparing Pre-discharge and posT-discharge tReatment Initiation With LCZ696 in heArt Failure patieNtS With Reduced ejectIon-fracTion hospItalized for an Acute decOmpensation eveNt (ADHF)
Brief Title: Comparison of Pre- and Post-discharge Initiation of LCZ696 Therapy in HFrEF Patients After an Acute Decompensation Event
Acronym: TRANSITION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CLCZ696B2401; 2015-003266-87 (EudraCT Number)
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Results first posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Acute decompensated heart failure; Reduced ejection fraction; Pre-discharge treatment; Post-discharge treatment; Angiotensin receptor neprilysine inhibitor; HFrEF
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pre-discharge treatment initiation (Other): Patients received first dose at any point after Randomization but no later than 12 h before discharge.
  Interventions: Drug: LCZ696
- Post-discharge treatment initiation (Other): Patients received first dose after discharge and up to 14 days thereafter.
  Interventions: Drug: LCZ696

INTERVENTIONS:
Drug: LCZ696 — LCZ696 film-coated tables were supplied to the investigators. Tablets were taken with a glass of water, and were administered with or without food.
  The target dose of LCZ696 was 200 mg twice daily. Starting dose of LCZ696 was either 50 or 100 mg, twice daily. The dose of LCZ696 should be doubled every 2-4 weeks to achieve the target dose of 200 mg twice daily, as tolerated by the patient.

SUMMARY:
To explore two modalities of treatment initiation (Pre-discharge, and Post-discharge) with LCZ696 in HFrEF patients following stabilization after an ADHF episode.

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalized due to acute decompensated HF episode (ADHF) as primary diagnosis) and consistent Signs & Symptoms
2. Diagnosis of HF New York Heart Association class II-to-IV and reduced ejection fraction: Left ventricular ejection fraction ≤ 40% at Screening
3. Patients did not receive any IV vasodilators (except nitrates), and/or any IV inotropic therapy from the time of presentation for ADHF to Randomization
4. Stabilized (while in the hospital) for at least 24 hours leading to Randomization.
5. Meeting one of the following criteria:

   * Patients on any dose of ACEI or ARB at screening
   * ACEI/ARB naïve patients and patients not on ACEI or ARB for at least 4 weeks before screening.

Exclusion Criteria:

1. History of hypersensitivity to the sacubitril, valsartan, or any ARBs, NEP inhibitors or to any of the LCZ696 excipients.
2. Symptomatic hypotension and/or a SBP below 110 mm Hg or SBP above 180 mm Hg prior to randomization
3. End stage renal disease at Screening; or estimated GFR below 30 mL/min/1.73 m2 (as measured by MDRD formula at Randomization.
4. Serum potassium above 5.4 mmol/L at Randomization.
5. Known history of hereditary or idiopathic angioedema or angioedema related to previous ACE inhibitor or ARB therapy
6. Severe hepatic impairment, biliary cirrhosis and cholestasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (137):
- Argentina (6):
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, Villa María, Córdoba Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Salta
  - Novartis Investigative Site, San Miguel de Tucumán
- Belgium (5):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Huy
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Ronse
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Czechia (13):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Karlovy Vary, Czech Republic
  - Novartis Investigative Site, Liberec, Czech Republic
  - Novartis Investigative Site, Tábor, Czech Republic
  - Novartis Investigative Site, Třebíč, Czech Republic
  - Novartis Investigative Site, Beroun, CZE
  - Novartis Investigative Site, Ostrava, CZE
  - Novartis Investigative Site, Brno-Bohunice
  - Novartis Investigative Site, Jihlava
  - Novartis Investigative Site, Kolín
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Slaný
- France (6):
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tourcoing
  - Novartis Investigative Site, Valenciennes
- Germany (21):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Leverkusen, North Rhine-Westphalia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Koeln-Nippes
  - Novartis Investigative Site, Langen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mönchengladbach
  - Novartis Investigative Site, Neuwied
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Rüsselsheim am Main
  - Novartis Investigative Site, Witten
- Italy (4):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Milan
- Lebanon (4):
  - Novartis Investigative Site, El Chouf, LBN
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Saida
- Norway (4):
  - Novartis Investigative Site, Ålesund
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Grålum
  - Novartis Investigative Site, Lillehammer
- Poland (7):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Puławy
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
  - Novartis Investigative Site, Lodz, Łódź Voivodeship
- Portugal (9):
  - Novartis Investigative Site, Vila Real, Portuigal
  - Novartis Investigative Site, Amadora
  - Novartis Investigative Site, Aveiro
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Covilha
  - Novartis Investigative Site, Guimarães
  - Novartis Investigative Site, Leiria
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Russia (5):
  - Novartis Investigative Site, Gatchina
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
- Saudi Arabia (3):
  - Novartis Investigative Site, Dammam
  - Novartis Investigative Site, Jeddah
  - Novartis Investigative Site, Riyadh
- Slovakia (9):
  - Novartis Investigative Site, Dunajská Streda, Slovak Republic
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Liptovský Mikuláš, Slovak Republic
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Dolný Kubín
  - Novartis Investigative Site, Martin
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Rimavská Sobota
  - Novartis Investigative Site, Trnava
- Spain (12):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Sanlúcar de Barrameda, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Barcelona/ Cataluny/Espanya
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Olot, Girona
  - Novartis Investigative Site, Móstoles, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Jönköping
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Geneva
- Turkey (Türkiye) (6):
  - Novartis Investigative Site, Eskişehir, Meselik
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Sivas
- United Kingdom (16):
  - Novartis Investigative Site, Westcliff-on-Sea, Essex
  - Novartis Investigative Site, Basingstoke, Hampshire
  - Novartis Investigative Site, Ashford, Kent
  - Novartis Investigative Site, Bridgend, Mid Glamorgan
  - Novartis Investigative Site, Portadown, Nothern Ireland
  - Novartis Investigative Site, Sunderland, Tyne and Wear
  - Novartis Investigative Site, Blackpool
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Swindon
  - Novartis Investigative Site, York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Straburzynska-Migaj E, Senni M, Wachter R, Fonseca C, Witte KK, Mueller C, Lonn E, Butylin D, Noe A, Schwende H, Lawrence D, Suryawanshi B, Pascual-Figal D; of TRANSITION Investigators. Early Initiation of Sacubitril/Valsartan in Patients With Acute Heart Failure and Renal Dysfunction: An Analysis of the TRANSITION Study. J Card Fail. 2024 Mar;30(3):425-435. doi: 10.1016/j.cardfail.2023.08.021. Epub 2023 Sep 9. PMID 37678704
- [Derived] Pascual-Figal D, Wachter R, Senni M, Bao W, Noe A, Schwende H, Butylin D, Prescott MF; TRANSITION Investigators. NT-proBNP Response to Sacubitril/Valsartan in Hospitalized Heart Failure Patients With Reduced Ejection Fraction: TRANSITION Study. JACC Heart Fail. 2020 Oct;8(10):822-833. doi: 10.1016/j.jchf.2020.05.012. Epub 2020 Aug 12. PMID 32800508
- [Derived] Senni M, Wachter R, Witte KK, Straburzynska-Migaj E, Belohlavek J, Fonseca C, Mueller C, Lonn E, Chakrabarti A, Bao W, Noe A, Schwende H, Butylin D, Pascual-Figal D; TRANSITION Investigators. Initiation of sacubitril/valsartan shortly after hospitalisation for acutely decompensated heart failure in patients with newly diagnosed (de novo) heart failure: a subgroup analysis of the TRANSITION study. Eur J Heart Fail. 2020 Feb;22(2):303-312. doi: 10.1002/ejhf.1670. Epub 2019 Dec 9. PMID 31820537
- [Derived] Wachter R, Senni M, Belohlavek J, Straburzynska-Migaj E, Witte KK, Kobalava Z, Fonseca C, Goncalvesova E, Cavusoglu Y, Fernandez A, Chaaban S, Bohmer E, Pouleur AC, Mueller C, Tribouilloy C, Lonn E, A L Buraiki J, Gniot J, Mozheiko M, Lelonek M, Noe A, Schwende H, Bao W, Butylin D, Pascual-Figal D; TRANSITION Investigators. Initiation of sacubitril/valsartan in haemodynamically stabilised heart failure patients in hospital or early after discharge: primary results of the randomised TRANSITION study. Eur J Heart Fail. 2019 Aug;21(8):998-1007. doi: 10.1002/ejhf.1498. Epub 2019 May 27. PMID 31134724
- [Derived] Pascual-Figal D, Wachter R, Senni M, Belohlavek J, Noe A, Carr D, Butylin D. Rationale and design of TRANSITION: a randomized trial of pre-discharge vs. post-discharge initiation of sacubitril/valsartan. ESC Heart Fail. 2018 Apr;5(2):327-336. doi: 10.1002/ehf2.12246. Epub 2017 Dec 14. PMID 29239515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized to pre-discharge group or post-discharged group.
Pre-assignment Details: The study consisted of 3 Epochs: the Screening Epoch (from signing of informed consent form to randomization), the treatment epoch (10 weeks following randomization), and a 16 weeks Follow-up Epoch following treatment epoch.
Groups:
- LCZ696 Pre-discharge Treatment Initiation: Patients received first dose at any point after Randomization but no later than 12 h before discharge.
- LCZ696 Post-discharge Treatment Initiation: Patients received first dose after discharge and up to 14 days thereafter.
Period: Overall Study
Arm/Group | LCZ696 Pre-discharge Treatment Initiation | LCZ696 Post-discharge Treatment Initiation
Started (Randomized) | 500 | 502
Started 10 Weeks Treatment Epoch | 497 | 501
Completed 10 Weeks Treatment Epoch | 460 | 455
Completed (Completed 16 weeks follow-up epoch) | 425 | 419
Not Completed | 75 | 83
Not completed — Physician Decision | 12 | 15
Not completed — Lost to Follow-up | 1 | 4
Not completed — Protocol Deviation | 0 | 4
Not completed — Non-compliance with study treatment | 5 | 5
Not completed — Death | 21 | 15
Not completed — Adverse Event | 10 | 8
Not completed — Withdrawal by Subject | 15 | 19
Not completed — Did not enter follow-up epoch | 7 | 10
Not completed — Death - no study drug received | 1 | 2
Not completed — Mis-randomized (not in treatment epoch) | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 Pre-discharge Treatment Initiation | LCZ696 Post-discharge Treatment Initiation | Total
Number analyzed (Participants) | 500 | 502 | 1002
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (12.27) | 67.0 (11.67) | 66.8 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 125 | 251
  Male | 374 | 377 | 751
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 488 | 486 | 974
  Black | 5 | 8 | 13
  Asian | 7 | 3 | 10
  Native American | 0 | 1 | 1
  Pacific Islander | 0 | 1 | 1
  Other | 0 | 1 | 1
  Unknown | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving the Target Dose of LCZ696 200 mg Bid at 10 Weeks Post Randomization
Description: Percentage of patients achieving and maintaining LCZ696 200 mg bid for at least 2 weeks leading to Week 10
Time Frame: 10 weeks after Randomization
Population: Safety Population (SAF). The SAF consisted of all randomized subjects who received at least one dose of study drug with the exception of those patients who were inadvertently randomized into the study. Subjects were analyzed according to treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 Pre-discharge Treatment Initiation | LCZ696 Post-discharge Treatment Initiation
Number analyzed (Participants) | 493 | 489
Participants | 224 | 248
Statistical Analysis 1: Comparison: LCZ696 Pre-discharge Treatment Initiation vs LCZ696 Post-discharge Treatment Initiation; Test type: Superiority; p = 0.099, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.896, 95% CI 2-sided [0.786 to 1.021]

2. Secondary Outcome: Percentage of Patients Achieving and Maintaining Either LCZ696 100 mg and/or 200 mg Bid
Description: Percentage of patients achieving and maintaining either LCZ696 100 mg and/or 200 mg bid for at least 2 weeks leading to Week 10
Time Frame: 10 weeks after Randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 Pre-discharge Treatment Initiation | LCZ696 Post-discharge Treatment Initiation
Number analyzed (Participants) | 493 | 489
Participants | 306 | 335
Statistical Analysis 1: Comparison: LCZ696 Pre-discharge Treatment Initiation vs LCZ696 Post-discharge Treatment Initiation; Test type: Superiority; p = 0.034, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.906, 95% CI 2-sided [0.827 to 0.993]

3. Secondary Outcome: Percentage of Patients Achieving and Maintaining Any Dose of LCZ696
Description: Percentage of patients achieving any dose of LCZ696 for at least 2 weeks leading to 10 weeks of treatment
Time Frame: 10 weeks after Randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 Pre-discharge Treatment Initiation | LCZ696 Post-discharge Treatment Initiation
Number analyzed (Participants) | 493 | 489
Participants | 424 | 438
Statistical Analysis 1: Comparison: LCZ696 Pre-discharge Treatment Initiation vs LCZ696 Post-discharge Treatment Initiation; Test type: Superiority; p = 0.089, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.960, 95% CI 2-sided [0.916 to 1.006]

4. Secondary Outcome: Percentage of Patients Permanently Discontinued From Treatment
Description: Percentage of patients permanently discontinued from LCZ696 (1) up to week 10 due to AEs, and (2) up to week 26 due to any reasons
Time Frame: 10 weeks after Randomization AND 26 weeks after randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 Pre-discharge Treatment Initiation | LCZ696 Post-discharge Treatment Initiation
Number analyzed (Participants) | 493 | 489
Participants
  up to week 10 due to AEs | 36 | 24
  up to week 26 due to any reasons | 83 | 78

5. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from randomization until first treatment with LCZ696. The period from randomization to first treatment was up to 14 days.
  On-treatment deaths were collected from first treatment with LCZ696 until 26 weeks post randomization.
Time Frame: From randomization until 26 weeks after randomization
Population: Safety Population (SAF) and randomized patients who died prior to first dose of study drug. The SAF consisted of all randomized subjects who received at least one dose of study drug with the exception of those patients who were inadvertently randomized into the study. Subjects were analyzed according to treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 Pre-discharge Treatment Initiation | LCZ696 Post-discharge Treatment Initiation
Number analyzed (Participants) | 494 | 491
Participants
  Pre-treatment deaths | 1 | 2
  On-treatment deaths | 23 | 13
  All deaths | 24 | 15

ADVERSE EVENTS:
Time Frame: From start of treatment until 26 weeks after randomization
Description: Analysis is based on the Safety Population (SAF). It consists of all randomized patients who received at least one dose of study drug.
  Deaths not included in the SAF (i.e. did not receive study drug) are presented separately in the Participant Flow and .
  Patients are analyzed according to treatment actually received.
Groups:
- Pre-discharge: Pre-discharge
- Post-discharge: Post-discharge
- All Patients: All patients
Arm/Group | Pre-discharge | Post-discharge | All Patients
All-Cause Mortality (participants affected / at risk) | 23/493 | 13/489 | 36/982
Serious Adverse Events (participants affected / at risk) | 159/493 | 134/489 | 293/982
Other Adverse Events (participants affected / at risk) | 200/493 | 201/489 | 401/982
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-discharge (N=493) | Post-discharge (N=489) | All Patients (N=982)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 5
Hypocoagulable state (Blood and lymphatic system disorders) | 1 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 2 | 3
Acute myocardial infarction (Cardiac disorders) | 1 | 3 | 4
Angina pectoris (Cardiac disorders) | 2 | 1 | 3
Angina unstable (Cardiac disorders) | 3 | 0 | 3
Arrhythmia (Cardiac disorders) | 2 | 1 | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 4 | 5 | 9
Atrial flutter (Cardiac disorders) | 1 | 1 | 2
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 2 | 2 | 4
Bradycardia (Cardiac disorders) | 2 | 1 | 3
Cardiac arrest (Cardiac disorders) | 4 | 1 | 5
Cardiac failure (Cardiac disorders) | 46 | 45 | 91
Cardiac failure acute (Cardiac disorders) | 11 | 9 | 20
Cardiac failure chronic (Cardiac disorders) | 3 | 2 | 5
Cardiac failure congestive (Cardiac disorders) | 1 | 4 | 5
Cardio-respiratory arrest (Cardiac disorders) | 1 | 2 | 3
Cardiogenic shock (Cardiac disorders) | 1 | 5 | 6
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 2 | 2
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 1
Left ventricular failure (Cardiac disorders) | 1 | 1 | 2
Low cardiac output syndrome (Cardiac disorders) | 1 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 1
Myocardial fibrosis (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 2
Myocardial ischaemia (Cardiac disorders) | 2 | 0 | 2
Palpitations (Cardiac disorders) | 1 | 0 | 1
Sinus arrest (Cardiac disorders) | 1 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 2 | 3
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 2 | 3
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 1 | 2
Ventricular tachycardia (Cardiac disorders) | 3 | 2 | 5
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 3
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2
Subileus (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 1
Impaired healing (General disorders) | 1 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 2
Non-cardiac chest pain (General disorders) | 2 | 5 | 7
Oedema peripheral (General disorders) | 1 | 3 | 4
Pyrexia (General disorders) | 0 | 1 | 1
Sudden cardiac death (General disorders) | 1 | 0 | 1
Sudden death (General disorders) | 2 | 0 | 2
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1 | 1
Biliary sepsis (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 4 | 5
Catheter site abscess (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 2
Device related infection (Infections and infestations) | 1 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1 | 1
Epididymitis (Infections and infestations) | 0 | 1 | 1
Erysipelas (Infections and infestations) | 1 | 3 | 4
Gangrene (Infections and infestations) | 1 | 1 | 2
Gastroenteritis (Infections and infestations) | 1 | 3 | 4
Influenza (Infections and infestations) | 1 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 7 | 8 | 15
Postoperative wound infection (Infections and infestations) | 1 | 0 | 1
Q fever (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 4 | 4
Sepsis (Infections and infestations) | 2 | 1 | 3
Septic phlebitis (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 1 | 2 | 3
Tuberculosis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 4 | 2 | 6
Urosepsis (Infections and infestations) | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 2 | 3
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Transplant failure (Injury, poisoning and procedural complications) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 2 | 0 | 2
Cardiac output decreased (Investigations) | 1 | 0 | 1
Ejection fraction abnormal (Investigations) | 1 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 2 | 2
General physical condition abnormal (Investigations) | 1 | 0 | 1
Heart rate abnormal (Investigations) | 1 | 0 | 1
Hepatic enzyme abnormal (Investigations) | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 6 | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Aphasia (Nervous system disorders) | 1 | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0 | 1
Brain injury (Nervous system disorders) | 1 | 0 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 2 | 3
Cognitive disorder (Nervous system disorders) | 1 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 2
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 2 | 2
Loss of consciousness (Nervous system disorders) | 0 | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 3 | 3 | 6
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1
Device battery issue (Product Issues) | 0 | 1 | 1
Device dislocation (Product Issues) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 12 | 7 | 19
Chronic kidney disease (Renal and urinary disorders) | 3 | 2 | 5
Haematuria (Renal and urinary disorders) | 0 | 2 | 2
Renal failure (Renal and urinary disorders) | 3 | 4 | 7
Renal impairment (Renal and urinary disorders) | 0 | 4 | 4
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 10
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 6 | 2 | 8
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 2 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-discharge (N=493) | Post-discharge (N=489) | All Patients (N=982)
Diarrhoea (Gastrointestinal disorders) | 17 | 29 | 46
Oedema peripheral (General disorders) | 20 | 26 | 46
Urinary tract infection (Infections and infestations) | 29 | 19 | 48
Hyperkalaemia (Metabolism and nutrition disorders) | 67 | 59 | 126
Dizziness (Nervous system disorders) | 32 | 30 | 62
Renal impairment (Renal and urinary disorders) | 36 | 24 | 60
Hypotension (Vascular disorders) | 71 | 67 | 138

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT02661217/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT02661217/SAP_001.pdf